CLINICAL TRIAL: NCT03121105
Title: A Pathologic-MRI Reappraisal of Patients With Atypical Idiopathic Inflammatory Demyelinating Disorders
Brief Title: Pathologic-MRI Findings in Atypical IIDD
Acronym: IIDD
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University Hospital, Strasbourg, France (Other); Rennes University Hospital (Other); University Hospital, Bordeaux (Other); University Hospital, Limoges (Other); Hospices Civils de Lyon (Other); Centre Hospitalier Universitaire de Nīmes (Other); Colmar Hospital (Unknown); Centre hospitalier de Perpignan (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0078
Record Dates: First submitted 2017-03-08; First posted 2017-04-19 (Actual); Last update posted 2018-05-07 (Actual); Status verified 2017-03

CONDITIONS: Idiopathic Inflammatory Demyelinating Disorders of the Central Nervous System
Keywords: Idiopathic Inflammatory demyelinating disorders of the central nervous system; Multiple Sclerosis; Neuromyelitis Optica; MRI; pahtological
MeSH Terms: conditions — Multiple Sclerosis; Neuromyelitis Optica

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our objective is to describe the pathologic and MRI findings in a series of patients with presumed demyelinating lesion of the central nervous system.

DETAILED DESCRIPTION:
Idiopathic inflammatory demyelinating disorders (IIDD) are a group of diseases with distinct clinical and magnetic resonnance imaging (MRI) features, the most frequent being Multiple Sclerosis (MS). MS can present with atypical MRI features that can be misleading. Neuromyelitis Optica Spectrum Disorder (NMOSD) is the main differential diagnosis. It has been demonstrated that some patient with NMOSD can also present with brain lesion that is sometimes difficult to diagnose. In this context, a retrospective series identifies 18 patients with centreal nervous system atypical demyelination and 1) pathological evidence of astrocytopathy and 2) immunohistochemistry demonstrating decrease of aqp4 binding. The aim of the study is to describe the radiological and pathological characteristics of a series of patients with pathologicaly proven atypical demyelination that underwent biopsy for diagnostic uncertainties.

This is a retrospective multicenter study. Inclusion criteria are: 1) Acute or subacute onset of neurological deficit, 2) Brain biopsy performed for diagnostic uncertainties revealing an active demyelinating lesion, 3) no known diagnosis of MS or NMOSD at the time of the biopsy and 4) no alternative diagnosis identified during the disease course.

All the medical records of the patients will be reviewed and the following data will be recorded: previous medical history including previous neurologic relapses, gender, age at onset, clinical symptoms at onset and diagnosis at last follow-up according to current diagnosis criteria for MS and NMOSD.

Brain MRI scanners will be analysed. The investigators will mainly focus on T1-, T2-, T2 gradient echo-, fluid- attenuated inversion recovery- and diffusion-weighted images. The following data will be recorded: number of lesions, location (cortical, juxtacortical, juxtaventricular, corpus callosum involvement, posterior fossa involvement), presence of a peripheral hyperintense/hypointense rim (on T2 sequence), and type of gadolinium enhancement (peripheral open or closed ring, central homogeneous or heterogeneous). The presence of oedema will be recorded and mass effect will be analysed. According to the classification of atypical demyelinating lesions (MAGNIMS group), patients will be classified as having either infiltrative, megacystic, balo-like, ring-like lesions or unclassified. Three neuropathologists (BL, BL and VR) blinded to the MRI and clinical datas will perform all the pathologic evaluations. Paraffin-embedded sections have been stained using hematoxylin & eosin, Luxol fast blue. Primary antibodies specific fot GFAP, CD3, CD8, CD20 and CD68 were used in routine practice. Additional immunohistochemical studies will be done using primary antiobodies specific for IgG and Aquaporin-4. The investigators will specifically look at the presence of 1) morphologic features suggestive of either MS (Creutzfeldt cells) or NMOSD (dystrophic astrocytes, myelin vacuolation, vascular hyalinization) 2) negative aquaporin-4 staining (suggestive of NMOSD) and 3) macrophages containing GFAP positive or Luxol fast blue positive debris.

ELIGIBILITY:
Inclusion Criteria:

* Presence of brain lesion in MRI suggestive of demyelinating lesions
* Biopsy analysis revealed active inflammation with active demyelination
* No known diagnosis of MS or Devic's disease or other diagnosis

Exclusion Criteria:

- NO

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 25 patients with cerebral MRI lesions suggestive of demyelinating lesions
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
pathological | 1 day
  pathological results: morphologic changes and specific immunostaining

SECONDARY OUTCOMES:
MRI (magnetic resonnance Imaging) | 1 day
  MRI results: characteristics of the MRI lesions

CONTACTS AND LOCATIONS:
Overall Officials: xavier AYRIGNAC, MD, Study Director — University Hospital, Montpellier

IPD SHARING:
Plan to Share IPD: Undecided
NC